CLINICAL TRIAL: NCT06964815
Title: Silibinin in Association With Concomitant Chemoradiotherapy and Maintenance Temozolomide in STAT3 Positive IDH Wild-type, Newly Diagnosed Glioblastoma Patients: a Multicenter, Double-blind, Placebo-controlled, Randomized Study
Brief Title: Silibinin in Association With Concomitant Chemoradiotherapy and Maintenance Temozolomide in STAT3 Positive IDH Wild-type, Newly Diagnosed Glioblastoma Patients
Acronym: STRONG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-GB-01-2024-STRONG
Record Dates: First submitted 2025-04-16; First posted 2025-05-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma; IDH Wild-type and STAT3-positive Glioblastoma
Keywords: Glioblastoma; IDH wild-type and STAT3-positive glioblastoma; silibinin; temozolomide; placebo
MeSH Terms: conditions — Glioblastoma | interventions — Silybin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silbrain_Experimental Arm (Experimental): Concomitant radiotherapy (60 gy in 30 fractions) + temozolomide 75mg/mq + silibinin 2 sachets/day dissolved in water throughout concomitant treatment followed by temozolomide cp, 150 mg/m2-200mg/m2, g1-5 q28d + silibinin 2 sachets/day dissolved in water, day 1-28, q28d for 6cycles. Silibinin will be continued until disease progression or up to 24 months. In patients who develop progression during temozolomide treatment, administration of silibinin will be continued for up to 6 months after the last dose of temozolomide.
  Interventions: Dietary Supplement: Silibinin as STAT3 inhibitor
- Placebo_Control Arm (Placebo Comparator): Concomitant radiotherapy (60 gy in 30 fractions) + temozolomide 75mg/mq + placebo 2 sachets/day dissolved in water throughout concomitant treatment followed by temozolomide cp, 150 mg/m2-200mg/m2, g1-5 q28d + placebo 2 sachets/day dissolved in water, day 1-28, q28d for 6 cycles. Silibinin/Placebo may be continued until disease progression at the discretion of the physician. Silibinin/Placebo will be continued until disease progression or up to 24 months. In patients who develop progression during temozolomide treatment, administration of silibinin (or placebo) will be continued for up to 6 months after the last dose of temozolomide.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Silibinin as STAT3 inhibitor — Sillbrain will be available as granulate in sachets of 3.7g and it will be administered twice a day during chemo-radiotherapy and day 1-28 in maintenance phase every cycle. Each 3.7 g sachet of Sillbrain contains 500 mg silibinin. Every patient will assume 2 sachets/day for a total of 1 g/day of silibinin.
  Arms: Silbrain_Experimental Arm
Other: Placebo — Placebo will be available as granulate in sachets of 3.7g and it will be administered twice a day during chemo-radiotherapy and day 1-28 in maintenance phase every cycle. Every patient will assume 2 sachets/day for a total of 1 g/day of placebo.
  Arms: Placebo_Control Arm

SUMMARY:
Multicenter, double-blind, placebo-controlled, randomized trial.

Patients affected by STAT3 positive newly diagnosed glioblastoma will be eligible. Patients are randomized using a stratified block randomization method with a 1:1 ratio in two arms:

• Experimental/Control arm: Concomitant radiotherapy (60 gy in 30 fractions) + temozolomide 75mg/mq + silibinin/placebo 2 sachets/day dissolved in water throughout concomitant treatment followed by temozolomide cp, 150 mg/m2-200mg/m2, g1-5 q28d + silibinin/placebo 2 sachets/day dissolved in water, day 1-28, q28d for 6-12 cycles. Silibinin/Placebo may be continued until disease progression at the discretion of the physician.

Patients will be stratified based on:

* Type of surgery (complete Vs partial)
* MGMT methylation status (methylated Vs non-methylated)
* ECOG PS (0-1 Vs 2)

ELIGIBILITY:
Inclusion Criteria:

* New histologically confirmed diagnosis of glioblastoma (WHO 2021)
* Local availability of MGMT methylation status
* Immunohistochemical positivity of activated STAT3 (pSTAT3) expression on the tumor tissue sample. STAT3 expression will be evaluated centrally by UOC Anatomia Patologica of Azienda Ospedale Università di Padova.
* Chemoradiotherapy start within 7 weeks from surgery
* Patients without disease progression after surgery
* Availability of paraffin-embedded tumor tissue
* Age ≥18 years
* ECOG PS 0-2; Karnofsky 100-70
* Signing of informed consent prior to any study procedure
* Patients (both males and females) should employ adequate contraceptive measures, which should be maintained during the whole duration of the trial (from screening to 6 months after the last dose of Temozolomide).
* Have adequate bone marrow, liver and kidney function, as measured by the following laboratory assessments conducted within 10 days before the start of study treatment:
* Hemoglobin > 9.0 g/dl
* Absolute neutrophil count (ANC) ≥1500/mm3 without granulocyte colony-stimulating factor (G-CSF) and other hematopoietic growth factors
* Platelet count ≥100,000/μl
* WBC ≥3.0 x 10 9 /L
* Total bilirubin <1.5 times the upper limit of normal
* ALT and AST <3 x the upper limit of normal
* Serum creatinine <1.5 times the upper limit of normal
* Glomerular filtration rate ≥ 30 mL/min/1.73 m2 according to the abbreviated formula Modified Diet in Renal Disease
* Alkaline phosphatase <2.5 x ULN
* PT-INR/PTT <1.5 x upper limit of normal (patients who are therapeutically anticoagulated with anticoagulant drugs will be able to participate provided there is no history of abnormal background in these parameters, based on history).
* Complete urinalysis
* Stable and decreasing corticosteroid dosage in the last 10 days before brain MRI

Exclusion Criteria:

* Patients diagnosed with glioblastoma (WHO grade IV 2021) who have only had a diagnostic biopsy
* Chemotherapy, immunotherapy, or antineoplastic therapy for glioblastoma
* Negative immunohistochemistry of STAT3 expression on the tumor tissue sample
* Diagnosis of another tumor or secondary brain localization
* In the investigator's judgment, any evidence of severe or uncontrolled systemic disease including: uncontrolled hypertension; hemorrhagic diathesis; active infection with HBV, HCV, HIV. Screening for such chronic conditions is not required by the protocol; bone marrow reserve or organ dysfunction as demonstrated by laboratory tests.
* Patients who are unable to comply with study procedures and requirements.
* Contraindication to Brain MRI
* Pregnant or breastfeeding patients
* Patients who are unable to swallow capsules or sachets dissolved in water.
* Patient unable to sign the Informed Consent
* Glioblastoma leptomeningeal dissemination
* Congestive heart failure classified as New York Heart Association (NYHA) Class 2 or higher; Unstable angina (symptoms of angina at rest) or new onset angina ≤3 months prior to screening; myocardial infarction <6 months prior to 'start of study treatment; cardiac arrhythmias requiring antiarrhythmic therapy, with the exception of beta-blockers or digoxin; uncontrolled hypertension (systolic blood pressure [SBP]>140 mmHg or diastolic blood pressure [DBP] >90 mmHg) despite optimal medical management.
* Arterial thrombotic or embolic events such as stroke and/or transient ischemic attacks) or
* Pulmonary embolism in the 6 months prior to the start of study treatment
* Ongoing infection with grade 2 or higher severity (NCI-CTCAE v 5.0)
* Known history of human immunodeficiency virus (HIV) infection; hepatitis B or C active or chronic requiring treatment with antiviral therapy
* History of organ allotransplantation
* Evidence or history of any bleeding diathesis (including mild hemophilia), regardless of its severity;
* Injuries, ulcers or bone fractures that have not fully resolved.
* Renal failure requiring hemodialysis or peritoneal dialysis
* Presenting interstitial lung disease with ongoing signs and symptoms at the time informed consent is obtained.
* Persistent proteinuria >3.5 g/24 hours as measured by urinary protein-creatinine ratio from a urine sample (≥ Grade 3, NCI-CTCAE v 5.0). CTCAE 5.0 is also available in Appendix 1.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Through study completion, an average of 2 years
  Evaluation of Progression Free Survival (PFS) in patients with newly diagnosed IDH wild-type and STAT3-positive glioblastoma using silibinin 2 sachets per day (1g/day), during chemoradiotherapy and maintenance treatment with temozolomide, compared with placebo. The progression free survival (PFS) will be determined as the time from the date of randomization to the date of disease progression determined using RANO 2.0 criteria or to the date of death, whichever occurs first. Patients without a PFS event at the time of analysis will be censored at the date of last assessment.

SECONDARY OUTCOMES:
Liver Toxicity | Through study completion, an average of 2 years
  Evaluation of liver toxicity. Assessment of liver toxicity will be derived from the assay of alanine aminotransferase (ALT) weekly during concomitant radio-chemotherapy treatment and monthly during maintenance temozolomide treatment, using the CTCAE v5.0 system to determine the degree of toxicity
Liver Toxicity | Through study completion, an average of 2 years
  Evaluation of liver toxicity. Assessment of liver toxicity will be derived from the assay of total and direct blood bilirubin weekly during concomitant radio-chemotherapy treatment and monthly during maintenance temozolomide treatment, using the CTCAE v5.0 system to determine the degree of toxicity
Liver Toxicity | Through study completion, an average of 2 years
  Evaluation of liver toxicity. Assessment of liver toxicity will be derived from the assay of aspartate aminotransferase (AST) weekly during concomitant radio-chemotherapy treatment and monthly during maintenance temozolomide treatment, using the CTCAE v5.0 system to determine the degree of toxicity
6/9-months Progression Free Survival (6/9m-PFS) | Through study completion, an average of 2 years
  Evaluation of 6/9-months Progression Free Survival (6/9m-PFS). The progression free survival at 6/9 months (6/9m-PFS) will be determined as the percentage of patient with progression of disease at 6 and 9 months
Objective Response Rate (ORR) | Through study completion, an average of 2 years
  Evaluation of Objective Response Rate (ORR). The objective response rate (ORR) will be defined as the percentage of patients with complete response (CR) and partial response (PR) determined using modified RANO criteria
EORTC QLQ-C30_Quality of Life | Through study completion, an average of 2 years
  Evaluation of Quality of Life assessed by EORTC QLQ-C30. EORTC QLQ-C30 has robust psychometric properties resulting from their use in several international cancer clinical trials. The EORTC QLQ-C30 (Aaronson et al, 1988) is a core measure designed to be supplemented with the disease specific module.
QLQ-BN20_Quality of Life | Through study completion, an average of 2 years
  Evaluation of Quality of Life assessed by QLQ-BN20. QLQBN20 has robust psychometric properties resulting from their use in several international cancer clinical trials.

CONTACTS AND LOCATIONS:
Locations (16):
- Italy (16):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, BO
  - IRST Dino Amadori, Meldola, FC
  - Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco ", Catania, Italia/Catania
  - Azienda Ospedaliera Universitaria - Careggi, Florence, Italia/FI
  - ARNAS G.Brotzu P.O Armando Businco, Cagliari, Italy/Cagliari
  - USL Nord Ovest Toscana - Livorno, Livorno, Italy/Livorno
  - Ospedale del Mare, ASL Napoli1 Centro, Napoli, italy/Napoli
  - Istituto Oncologico Veneto, Padua, Italy/Padova
  - Istituto Neurologico Nazionale a Carattere Scientifico IRCCS - Fondazione Mondino, Pavia, Italy/Pavia
  - Azienda Ospedaliera Universitaria G.Martino, Messina, ME
  - Istituto Tumori Regina Elena IRCCS, Roma, RM
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - Policlinico San Martino - Genova, Genova
  - Ospedale A. Manzoni Lecco, Lecco
  - Humanitas Cancer Center, Milan
  - IRCCS Ospedale Galeazzi Sant'Ambrogio, Milan

IPD SHARING:
Plan to Share IPD: Undecided